

# **Clinical Development**

# ABL001/ASCIMINIB

#### CABL001AUS04 / NCT04666259

An open label, multi-center Phase IIIb study of asciminib (ABL001) monotherapy in previously treated patients with chronic myeloid leukemia in chronic phase (CML-CP) with and without T315I mutation (AIM4CML)

# **Statistical Analysis Plan (SAP)**

Document type: SAP Documentation

Document status: Amendment 2.0

Release date: 16-Feb-2024

Number of pages: 42

Template version 4.0, Effective from 23-Apr-2021

# **Document History – Changes compared to previous final version of SAP**

| Date | Time point | Reason for update | Outcome for update | Section and<br>title impacted<br>(Current) |
|---|---|---|---|---|
| 06- Apr- 2021 | Prior to DB First Patient First Visit | Creation of final version | N/A - First version | NA |

Creation of Prior to DB lock 13- Jan- 2023 Amendment 1.0 of primary analysis

Replaced 'sequentially' allocated with 'randomly' allocated in all instances

All sections

Removed the note on cut-ff date for primary analysis

Section 2.1

Removed week 60 assessment and updated time interval for week 72 in table for molecular assessment

Added statement for mapping EOT assessment

Added week 72 for hematologic response assessment



Updated the criteria for generating TFLs for subgroup analysis

Section 2.2.1

Replaced duration of exposure with non-zero dose with Time on treatment

Section 2.4.1

Deleted cardiovascular risk factors not mentioned in Ecrf

Section 2.6.5.3

Deleted section on liver function risk assessment as the data is not collected

Updated the secondary objectives to align with Section 2.8

protocol

Updated the criteria to handle missing MMR rates Section 2.8.3



15- Feb- 2024 Prior to DB lock Creation of Amendment 2.0 of Interim analysis

# **Table of contents**

| Table | of contents | s | 5 |
|---|---|---|---|
| l Introduc | tion | | 11 |
| 1.1 | Study de | esign | 11 |
| 1.2 | Study of | bjectives and endpoints | 13 |
| 2 Statistica | al methods. | | 14 |
| 2.1 D | ata analysis | s general information | 14 |
| | 2.1.1 Ge | eneral definitions | 15 |
| 2.2 | Analysis | s sets | 19 |
| | 2.2.1 | Subgroup analyses | 19 |
| 2.3 | Patient of | disposition, demographics, and other baseline characteristics | 20 |
| | 2.3.1 De | emographics and baseline characteristics | 20 |
| | 2.3.2 Di | agnosis and extent of cancer - CML | 20 |
| | 2.3.3 Me | edical history | 20 |
| | 2.3.4 Pa | tient disposition | 21 |
| | 2.3.5 Pro | otocol deviations | 21 |
| 2.4 | Treatme | ents (study medication, rescue medication, concomitant therapies, compliance) | 22 |
| | 2.4.1 | Duration of exposure to study medication | 22 |
| | 2.4.2 | Prior, concomitant and post therapies/medication | 23 |
| 2.5 | Analysis | s of the primary objective | 24 |
| | 2.5.1 | Primary endpoint | 25 |
| | 2.5.2 | Statistical hypothesis, model, and method of analysis | 25 |
| | 2.5.3 | Handling of missing values | 25 |
| 2.6 | Safety a | nalyses | 25 |
| | 2.6.1 | Adverse events (AEs) | 25 |
| | 2.6.2 | Adverse events of special interest / grouping of AEs | |
| | 2.6.3 | Deaths | 26 |
| | 2.6.4 | Laboratory data | 26 |
| | 2.6.5 | Other safety data | 27 |
| 2.7 A | nalysis of t | he key secondary objective | 28 |
| 2.8 A | nalysis of t | he secondary objective(s) | 28 |
| | 2.8.1 Se | condary safety endpoints | 29 |
| | | econdary efficacy endpoints | |
| | | andling of missing values/censoring/discontinuations | |
| <u></u> _ | 2.8.4 Sta | atistical hypothesis, model, and method of analysis | |
| | | | 32 |
| | | | 33 |
| | | | 34 |

| | | | | 35 |
|---|---|---|---|---|
| | 2.10 I | nterim ana | alysis | 35 |
| 3 | Samp | le size calo | culation | 35 |
| 4 | Chang | ge to proto | ocol specified analyses | 36 |
| 5 | Appe | ndix | | 36 |
| | 5.1 | Imputat | tion rules | 36 |
| | | 5.1.1 | Study drug | 36 |
| | | 5.1.2 | AE, ConMeds and safety assessment date imputation | 36 |
| | 5.2 | AEs coo | ding/grading | 38 |
| | 5.3 | Laborat | tory parameters derivations | 38 |
| | | 5.3.1 D | rerivation of PCR results and loss of response(s) | 39 |
| | 5.4 | Listing | of AESIs | 41 |
| 6 | Refer | ence | | 42 |

# List of abbreviations

| ADME Absorption, Distribution, Metabolism, and Excretion AE Adverse Event AESI Adverse event of special interest ALP Alkaline phosphatase ALT Alanine aminotransferase/glutamic pyruvic transaminase/GPT ANC Absolute neutrophil count AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | ABL | Abelson proto-oncogene |
|---|---|---|
| AESI Adverse event of special interest ALP Alkaline phosphatase ALT Alanine aminotransferase/glutamic pyruvic transaminase/GPT ANC Absolute neutrophil count AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | ADME | Absorption, Distribution, Metabolism, and Excretion |
| ALP Alkaline phosphatase ALT Alanine aminotransferase/glutamic pyruvic transaminase/GPT ANC Absolute neutrophil count AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | AE | Adverse Event |
| ALP Alkaline phosphatase ALT Alanine aminotransferase/glutamic pyruvic transaminase/GPT ANC Absolute neutrophil count AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | AESI | Adverse event of special interest |
| ANC Absolute neutrophil count AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | ALP | |
| AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | ALT | Alanine aminotransferase/glutamic pyruvic transaminase/GPT |
| ATP Adenosine triphosphate AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | ANC | Absolute neutrophil count |
| AUC Area under the curve AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | AST | Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT |
| AV block Atrioventricular block b.i.d. bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | 1 1 |
| bis in die/twice a day BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML-AP Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | AUC | Area under the curve |
| BC Blast crisis BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | block Atrioventricular block |
| BCR Breakpoint Cluster Region gene BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | · |
| BCR-ABL BCR-ABL fusion gene (also called the Philadelphia chromosome) BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| BID bis in diem/twice a day BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| BMI Body Mass Index CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| CBC Complete Blood Count CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| CDP Clinical Development Plan CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| CDS Core Data Sheet CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CBC | Complete Blood Count |
| CHR Complete Hematological Response CI Confidence Interval CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CDP | Clinical Development Plan |
| CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CDS | Core Data Sheet |
| CK Creatinine Kinase CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CHR | Complete Hematological Response |
| CML Chronic Myelogenous Leukemia CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CI | Confidence Interval |
| CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CK | Creatinine Kinase |
| CML-AP Chronic Myelogenous Leukemia-Accelerated Phase CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| CMO&PS Chief Medical Office and Patient Safety CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CML | Chronic Myelogenous Leukemia |
| CO Country Organization CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CML-AP | Chronic Myelogenous Leukemia-Accelerated Phase |
| CO2 carbon dioxide CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CMO&PS | Chief Medical Office and Patient Safety |
| CP Chronic phase CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CO | Country Organization |
| CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | CO2 | carbon dioxide |
| CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | | |
| CRF Case Report/Record Form (paper or electronic) CRO Contract Research Organization | СР | Chronic phase |
| CRO Contract Research Organization | CRF | Case Report/Record Form (paper or electronic) |
| CCD CIT 1 1 1 1 | CRO | |
| USP Ulinical study protocol | CSP | Clinical study protocol |
| CSR Clinical study report | | • • • |
| CTCAE Common Terminology Criteria for Adverse Events | | |
| CV Coefficient of variation | | |

| Amendment | |
|---|---|
| CYP3A4 | Cytochrome P450 3A4 |
| DBP | Diastolic Blood Pressure |
| DDI | Drug-drug interaction |
| DLCO | Carbon monoxide diffusing capacity |
| DLT | Dose Limiting Toxicity |
| DMC | Data Monitoring Committee |
| DNA | Deoxyribonucleic acid |
| DQF | Data Query Form |
| DS&E | Drug Safety and Epidemiology |
| DSMB | Data Safety Monitoring Board |
| DSUR | Development safety update report |
| ECG | Electrocardiogram |
| eCOA | Electronic Clinical Outcome Assessment |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EDC | Electronic data capture |
| ELISA | Enzyme-linked immunosorbent assay |
| ELN | European Leukemia Network |
| EOT | End of Treatment |
| eSAE | Electronic Serious Adverse Event |
| eSource | Electronic Source |
| EU | European Union |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FIH | First In Human |
| FSH | Follicle Stimulating Hormone |
| GCP | Good Clinical Practice |
| GCS | Global Clinical Supply |
| GDPR | General Data Protection Regulation |
| GFR | Glomerular Filtration Rate |
| GGT | Gamma-glutamyl transferase |
| Н | Hour |
| hADME | Human ADME study (Absorption, Distribution, Metabolism and Excretion) |
| HBsAg | Hepatitis B surface antigen |
| HDL | High density lipoprotein |
| i.v. | Intravenous |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use |
| IEC | Independent Ethics Committee |
| INR | International normalized ratio |
| IWRS | Interactive Web Response System |
| IRB | Institutional Review Board |
| מאוו | Institutional Review Board |

| IRT | Interactive Response Technology that includes Interactive Voice Response |
|---|---|
| | System and |
| Km | Michaelis-Menten constant |
| K-M | Kaplan-Meyer |
| LDH | Lactate dehydrogenase |
| LDL | Low density lipoprotein |
| LFT | Liver function test |
| LLN | Lower limit of normal |
| LLOQ | lower limit of quantification |
| LSC | Leukemia stem cell |
| MCyR | Major Cytogenetic Response |
| mCyR | Minor Cytogenetic Response |
| MedDRA | Medical dictionary for regulatory activities |
| Mg | milligram(s) |
| mL | milliliter(s) |
| MMR | Major Molecular Response |
| MRI | Magnetic resonance imaging |
| NCDS | Novartis Clinical Data Standards |
| NOVDD | Novartis Data Dictionary |
| | , |
| OS | Overall survival |
| p.o. | oral(ly) |
| PCR | Polymerase Chain Reaction |
| PCyR | Partial Cytogenetic Response |
| PD | Pharmacodynamic(s) |
| Ph+ | Philadelphia chromosome positive |
| PHI | Protected Health Information |
| PLT | Platelets |
| PPD | Premature Participant Discontinuation |
| PPS | Per-protocol set |
| PSD | Premature Subject Discontinuation |
| PSUR | Periodic safety update report |
| PT | prothrombin time |
| QD | Quaque die/once a day |
| QMS | Quality Management System |
| QT | Q to T interval (ECG) |
| QTcF | QT interval corrected by Fridericia's formula |
| R Value | ALT/ALP x ULN |
| RAP | The Report and Analysis Plan |
| RBC | red blood cell(s) |
| TOC | 104 01004 0011(5) |

| i Amendinen | t 1.0 OABEUUTAU |
|---|---|
| RDC | Remote Data Capture |
| RDE | Recommended dose for expansion |
| REB | Research Ethics Board |
| RNA | Ribonucleic acid |
| RoW | Rest of World |
| RP2D | Recommended phase two dose |
| RQ-PCR | Real time quantitative polymerase chain reaction |
| s.c. | Subcutaneous |
| SAE | Serious Adverse Event |
| SAP | The Statistical Analysis Plan (SAP) is a regulatory document which provides evidence of preplanned analyses |
| SBP | Systolic Blood Pressure |
| SC | Steering committee |
| sCR | serum creatinine |
| SD | Standard deviation |
| SGOT | Serum glutamic oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SmPC | Summary of Product Characteristics |
| SOP | Standard Operating Procedure |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TBIL | Total bilirubin |
| TD | Study medication Discontinuation |
| TdP | Torsades de Pointes |
| TKI | Tyrosine Kinase Inhibitor |
| TTF | Time to treatment failure |
| UGT | Uridin diPhospho-glucuronosyltransferase |
| ULN | Upper limit of normal |
| ULQ | upper limit of quantification |
| US | United States |
| USPI | US prescribing information |
| UTI | Urinary Tract Infection |
| WBC | White blood cell(s) |
| WHO | World Health Organization |
| WoC | Withdrawal of Consent |

#### 1 Introduction

This statistical analysis plan (SAP) describes all planned analyses of primary objective, secondary objectives for the clinical study reports (CSR) of study CABL001AUS04, a phase 3b, multi-center, open-label, study of oral asciminib monotherapy in patients with Chronic Myelogenous Leukemia in chronic phase (CML-CP), previously treated with at least 2 ATP-site tyrosine kinase inhibitors (TKI) (i.e. imatinib, nilotinib, bosutinib, dasatinib or ponatinib) in case of absence of T315I mutation or previously treated with at least 1 ATP-site tyrosine kinase inhibitors (i.e. imatinib, nilotinib, bosutinib, dasatinib or ponatinib) in case of presence of T315I mutation.

The main purpose of this document is to describe the statistical methodology that will be used for this clinical study.

The analysis described here will be conducted by Novartis using statistical software SAS® Version 9.4 or higher, according to the Statistical methods and data analysis Section 12of the study protocol.

Unless otherwise specified, the statistical methodologies including the analysis sets, analysis models, algorithms and conventions are following the Oncology study protocol CABL001AUS04 version 03.

# 1.1 Study design

This study will be a multicenter Phase IIIb open-label, three-cohort study of asciminib in patients with CML-CP without T315I mutation who have had at least 2 prior TKIs and CML- CP harboring the T315I mutation with at least 1 prior TKI (Figure 1-1). Approximately 115 patients will be enrolled in the study. 90 patients without T315I mutation will be randomly selected in Cohort A & B (45 patients per Cohort). Remaining 25 patients with T315I mutation will be enrolled in Cohort C.

The study will contain following Cohorts:

- Cohort A (45): where patients will receive asciminib at 40 mg twice daily
- Cohort B (45): where patients will receive asciminib at 80 mg once daily
- Cohort C (25): patients harboring the T315I mutation will be treated on the dose of 200 mg twice daily.

Figure 1-1 Schematic of study design



For patients without T315I mutation, patients will be selected randomly between Cohort A, where patients will be given asciminib at 40 mg twice daily (BID) and Cohort B, where patients will receive asciminib at 80 mg daily (QD) to minimize selection bias. In Cohort C, patients harboring the T315I mutation will be enrolled and treated on the dose of 200 mg twice daily (BID). The higher dose required for that patient population is related to its required concentration to attain optimal blockade of the kinase activity. Patients will continue therapy until disease progression, unacceptable toxicity, or elective treatment discontinuation.

AEs, SAEs, and laboratory evaluation for 24 weeks is the primary endpoint in this study. AEs, SAEs and laboratory evaluation for Cohort A, B and Cohort C, during 48, 72 weeks is the secondary safety endpoint.

The primary analysis will be performed after all patients have been followed for at least 24 weeks or have discontinued study earlier. The end of study medication analysis will be performed after all patients have been followed for at least 72 weeks or have discontinued study earlier. The PFS/OS update analysis will be performed during 24, 48 and 72 weeks of the last patient received the first study dose.

No formal interim efficacy analysis is planned in this study. As the primary time point is by 24 weeks, the primary analysis will be an interim analysis performed when the last patient completes 24 weeks of treatment or discontinues early. As appropriate, annual interim analyses may be planned for publication or any regulatory purpose. Only summary statistics will be provided.

Final Analysis will be performed when the last patient completes 72 weeks of treatment or discontinues early.

# 1.2 Study objectives and endpoints

# Table 1-1 Objective(s) Endpoint(s)

| • To evaluate safety profile of monotherapy asciminib in CML- CP in 3L and beyond, for Cohorts A and B Secondary Objective(s) En | AEs, SAEs and laboratory evaluation for Weeks. |
|---|---|
| asciminib in CML- CP in 3L and beyond, for Cohorts A and B Secondary Objective(s) En | • |
| • To evaluate safety profile of monotherapy • A | ndpoint(s) for secondary objective(s) |
| asciminib in CML- CP in 3L and beyond, 24 for Cohort C | AEs, SAEs and laboratory evaluation for Weeks. |
| asciminib in CML- CP in all Cohorts A, B Co | AEs, SAEs and laboratory evaluation for ohort A, Cohort B and Cohort C, during 8, 72 weeks |
| <u> </u> | Rate of CHR, MR2, MMR, by 12, 24, 48, weeks of therapy |
| <u> </u> | Rate of MR4, MR4.5 by 48, 72 weeks of erapy |
| • To estimate time to hematologic and molecular response | Time to CHR, MR2, MMR, MR4, MR4.5 |
| | Duration of CHR, MR2, MMR, MR4 and R4.5 |
| • To Evaluate the progression free survival (PFS) | PFS during 24, 48 and 72 weeks |
| • To Evaluate Overall Survival (OS) • C | OS during 24, 48 and 72 weeks |

#### 2 Statistical methods

# 2.1 Data analysis general information

All analysis will be performed by Novartis.

It is planned that the data from all centers that participate in this protocol will be used for analysis. Analysis datasets and statistical outputs will be produced using the most recent SAS® Version 9.4 (SAS Institute Inc., Cary, NC, USA) or higher, and stored in Novartis global programming & statistical environment (GPS).

There is no formal planned interim analysis.

# Data included in the analyses

The analysis data cut-off dates for the planned analyses are:

- Primary analysis: After random allocation of all patients in their respective Cohort, have been on study medication for 24 weeks or discontinued earlier, i.e., LPFT + 24 weeks.
- Final safety, efficacy analyses: 30 days after all patients have been on treatment for at least 72 weeks or discontinued earlier, i.e., LPFT + 72 weeks + 30 days. (Note: After the study medication period, the assigned study medication will be made available, may be outside of this study, to patients who in the opinion of the investigators are still deriving clinical benefit.)

All statistical analyses will be performed using all data collected in the database up to the respective data cut-off date. All data with an assessment date or event start date (e.g., vital sign assessment date or start date of an adverse event) prior to or on the cut-off date will be included in the analysis. Any data collected beyond the cut-off date will not be included in the analysis and will not be used for any derivations.

All events with start date before or on the respective cut-off date and end date after the respective cut-off date will be reported as ongoing. The same rule will be applied to events starting before or on the respective cut-off date and not having documented end date. This approach applies, in particular, to adverse event and concomitant medication reports. For these events, the end date will not be imputed and therefore will not appear in the listings.

### General analysis conventions

**Pooling of centers:** Unless specified otherwise, data from all study centers will be pooled for the analysis. Due to expected small number of patients enrolled at centers, no center effect will be assessed.

Categorical data (e.g., gender, race, etc.) will be summarized by frequency and percentages by Cohort along with 95% Confidence interval (as appropriate); a missing category will be included as applicable. Percentages will be calculated using the number of patients in the relevant Cohort as the denominator. 95% Confidence Interval for the percentages will be evaluated using Clopper-pearson method.

Continuous data (e.g., age, body weight, etc.) will be summarized by appropriate descriptive statistics (i.e., mean, standard deviation, median, minimum, Q1, Q3, and maximum) by Cohort

estimated rate by specific timepoints will be reported along with their respective 95% Confidence interval(s).

#### 2.1.1 General definitions

#### Investigational drug and study medication

*Investigational drug* will refer to the ABL001 only. Whereas *study medication* will refer to ABL001 [asciminib (40 mg BID, 80 mg QD or 200 mg BID)]. Novartis is supplying asciminib to the investigational site as 20 mg and 40 mg tablets.

#### **Treatment Cohorts**

Patients without T315I mutation status are selected randomly between Cohort A (without T315I) and Cohort B (without T315I). Patients harboring the T315I mutation are allocated to Cohort C.

| Without T315 | I mutation | With T315I mutation |
|--------------|------------|---------------------|
| Cohort A | Cohort B | Cohort C |
| 40 mg BID | 80 mg QD | 200 mg BID |

# Date of first administration of study medication

The <u>date of first administration of study medication</u> is derived as the first date when a non-zero dose of study medication was administered as per the Dosage Administration Record (DAR) electronic case report form (eCRF). The date of first administration of study medication will also be referred as *start of study medication*.

The <u>date of first administration of study medication</u> is the same as the date of first administration of investigational drug.

# Date of last administration of study medication

The <u>date of last administration of study medication</u> is defined as the last date when a non-zero dose of study medication was administered as per the DAR eCRF.

The <u>date of last administration of study medication</u> is the same as the date of last administration of investigational drug.

#### Study day

The study day describes the day of the event or assessment date, relative to the reference start date.

- The date of the event (visit date, onset date of an event, assessment date, etc.) reference start date + 1 if event is on or after the reference start date;
- The date of the event (visit date, onset date of an event, assessment date, etc.) reference start date if event precedes the reference start date.

| The reference start date for safety asses | ssments (e.g., adverse | event onset, laboratory abnormality |
|---|---|---|
| occurrence, vital sign measurement, dose | interruption, etc. | ) is the start of study medication. |

The reference start date for all other, non-safety assessments (e.g., molecular response, survival time, disease progression, ECOG performance status, etc.) is the date of random allocation of patient to their respective Cohort.

The study day will be displayed in the data listings. If an event starts before the reference start date, the study day displayed on the listing will be negative.

For "time since event" data (e.g., medical history), the duration (in days) will be calculated as treatment start date-diagnosis date.

### Time unit

A year length is defined as 365.25 days. A month length is 30.4375 (=365.25/12) days. If duration is reported in months, duration in days will be divided by 30.4375. If duration is reported in years, duration in days will be divided by 365.25.

A week length is defined as 7 days. If duration is reported in weeks, duration in days will be evaluated by dividing duration in weeks by 7. All the time related study endpoints will be reported in Weeks, until stated or specified.

#### **Baseline**

For safety & efficacy evaluations, the last available assessment on or before the date of start of study medication of asciminib (40 mg BID, 80 mg QD & 200 mg BID) is taken as "baseline" assessment. For pre-dose electrocardiogram (ECG), the last available assessment before the treatment start date/time is used for baseline.

For ECGs, where study requires multiple replicates per time point, the average of these measurements would be calculated for baseline (if not already available in the database).

In rare cases where multiple laboratory measurements meet the baseline definition, with no further flag or label that can identify the chronological order, then the following rule should be applied: If values are from central and local laboratories, the value from central assessment should be considered as baseline.

If patients have no value as defined above, the baseline result will be missing.

#### On-treatment assessment/event and observation periods

For adverse event, reporting the overall observation period will be divided into two mutually exclusive segments:

- **Pre-treatment period**: from day of patient's informed consent to the day before first administration of study medication
- *On-treatment period*: from date of first administration of study medication to 30 days after date of last actual administration of any study medication (including start and stop date).

<u>Note:</u> Patients will be treated for up to LPFT + 72 weeks. This will be the last actual administration of study medication for each patient if the patient has not discontinued study medication earlier. After this period, the assigned study medication will be made available, may be outside of this study, to patients who in the opinion of the investigators are still deriving clinical benefit.

#### Visit window

#### Windows for multiple assessments

In order, to summarize molecular response, Hematologic Response, collected over time (including unscheduled visits), the assessments will be time slotted. The following general rule will be applied in creating the assessment windows: If more than one assessment is done within the same time window, the assessment performed closest to the target date will be used. If two assessments within a time window are equidistant from the target date, then the average of the two assessments will be used. If multiple assessments on the same date, then the average will be used. Data from all assessments (scheduled and unscheduled), including multiple assessments, will be listed.

Table 2-1 Time windows for molecular response (BCR-ABL1 quantification by RQ-PCR)

| Assessment | Target day of assessment | Time Interval |
|------------|--------------------------|--------------------|
| Baseline | ≤ 1 | ≤ Day 1# |
| Week 4 | 29 | Day 2 to day 57 |
| Week 12 | 85 | Day 58 to day 127 |
| Week 24 | 169 | Day 128 to day 211 |
| Week 36 | 253 | Day 212 to day 295 |
| Week 48 | 337 | Day 296 to day 421 |
| Week 72 | 505 | Day 422 to day 589 |

# Day 1 = Date of random allocation of patients

EOT assessments are mapped to the time points as needed.

 Table 2-2
 Time windows for Hematologic response assessment

| Assessment | Target day of assessment | Time Interval |
|------------|--------------------------|--------------------|
| Week 12 | 85 | Day 2 to day 127 |
| Week 24 | 169 | Day 128 to day 211 |
| Week 36 | 253 | Day 212 to day 295 |
| Week 48 | 337 | Day 296 to day 421 |
| Week 72 | 505 | Day 422 to day 589 |

# Day 1 = Date of random allocation of patients

EOT assessments are mapped to the time points as needed.



#### Last contact date

The last contact date will be derived for patients not known to have died at the respective analysis data cut-off date using the last complete date among the following:

Table 2-5 Last contact date data sources

| Source data | Conditions |
|---|---|
| Date of random allocation | No condition |
| Last contact date/last date patient was known to be alive from Survival Follow-up page | Patient status is reported to be alive, lost to follow-up or unknown |
| Start/End dates from further antineoplastic therapy | Non-missing medication/procedure term |
| Start/End dates from drug administration record | Non-missing dose. Doses of 0 are allowed |
| End of treatment date from end of treatment page | No condition |
| Any specific efficacy (molecular or cytogenetic) assessment date if available | Evaluation is marked as 'done' |
| Laboratory/ collection dates | Sample collection marked as 'done' |
| Vital signs date | At least one non-missing parameter value |
| Performance status date | Non-missing performance status |
| Start/End dates of AE | Non-missing verbatim term |

The last contact date is defined as the latest complete date from the above list on or before the respective data cut-off date. The cut-off date will not be used for last contact date unless the patient was seen or contacted on that date. No date post cut-off date will be used. Completely imputed dates (e.g., the analysis data cut-off date programmatically imputed to replace the missing end date of a dose administration record) will not be used to derive the last contact date.

The last contact date will be used for censoring of patients in the analysis of overall survival.

# 2.2 Analysis sets

# Full Analysis Set (FAS)

The Full Analysis Set (FAS) comprises all patients to whom study medication has been assigned. According to the intent to treat principle, patients will be analyzed according to the study medication and Cohort they have been assigned.

All the secondary efficacy endpoints will be analyzed using FAS.

# Safety Set (SS)

The **Safety Set (SS)** includes all patients who received at least one dose of study medication. Patients will be analyzed according to the study medication (regimen) they actually received.

The primary and all safety endpoints analysis will be performed on Safety Set.



#### **Patient Classification**

Patients may be excluded from the analysis populations defined above based on the protocol deviations entered in the database and/or on specific patient classification.

During the study, major and minor protocol deviations will be identified and collected on an ongoing basis as they occur. Refer to special data handling in data management documents. The decision whether patients will be included or excluded in the appropriate analysis sets will be determined based on the severity levels of the PDs.

# 2.2.1 Subgroup analyses

**Subgroup analyses** will be performed based on the patient's baseline status:

- Age:  $(< 65 \text{ years}; \ge 65 \text{ years})$
- Patients with resistance: (BCR-ABL ratio at baseline >10%)
- Previous treatment with Ponatinib (Yes or No)
- By number of prior TKI therapies:  $2, 3, \ge 4$

Summary tables and figures will be generated only for subgroups with at least 5% of the total sample size of full analyses set (for efficacy endpoint) or safety set (for safety endpoint).

All primary and secondary endpoints will be analyzed and summarized within each subgroup. Additionally, as the study is ongoing during COVID-19 pandemic, to address the impact of COVID-19 (if any) AEs, SAEs, Abnormal lab findings and notable vital signs will be summarized and reported if COVID-19 infected patient count exceeds 5% of the total sample size of safety set.

As appropriate, given the significance of the impact of COVID-19 on the enrolled patients, a sensitivity analysis may be performed on the safety and efficacy data evaluating the impact of COVID-19 on the study, if COVID-19 infected patient count exceeds 5% of the total sample size.

# 2.3 Patient disposition, demographics, and other baseline characteristics

# 2.3.1 Demographics and baseline characteristics

FAS will be used for all baseline and demographic summaries and listings unless otherwise specified. Patient demographics and baseline characteristics collected will include the following: date of birth, gender (and childbearing potential for female), race and ethnicity, height, weight, all relevant medical history including cardiovascular disease history, CML disease history, including mutation status, and prior and concomitant medication including prior TKI therapy and antineoplastic medication.

Physical examination including, extramedullary involvement, performance status, vital signs, ECGs, and laboratory assessments performed at screening will be summarized by Cohort.

Summaries will be reported for all patients. No inferential statistics will be provided.

All demographic and baseline disease characteristics data will be summarized by Cohort. Categorical data (e.g., age groups: < 65, and  $\ge 65$  years, sex, race, ethnicity, ECOG performance status) will be summarized by frequency counts and percentages; the number and percentage of patients with missing data will be provided. Continuous data (e.g., age, weight, height, body mass index) will be summarized by descriptive statistics (N, mean, median, standard deviation, minimum and maximum), where BMI (kg/m²) will be calculated as weight[kg] / (height[m]²) using weight at screening.

The number (%) of patients in each Cohort A, B & C ("With T315I Mutation" or "Without T315I Mutation") based on data obtained from the IRT system will be summarized based on their respective assigned cohort for all the patients in their respective analysis sets.

#### 2.3.2 Diagnosis and extent of cancer - CML

All diagnosis and extent of CML data will be summarized by Cohort. One summary table will include time (years) since initial diagnosis (descriptive statistics with N, mean, median, standard deviation, minimum and maximum) and historical mutation (frequency counts and percentages). Another table will include extramedullary involvement (frequency counts and percentages).

#### 2.3.3 Medical history

Significant findings that were present prior to the signing of informed consent will be included in the Relevant Medical History/Current Medical Conditions page on the patient's eCRF. Significant new findings that begin or worsen after informed consent will be recorded on the AE page of the patient's eCRF and will be summarized & listed overall and by Cohort.

Medical history and ongoing conditions, including toxicity grade entered on eCRF will be summarized and listed by Cohort. The summary will be presented by primary system organ class (SOC), preferred term (PT) and Cohort. Medical history and current medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) terminology. The MedDRA version used for reporting will be specified in the CSR and as a footnote in the applicable tables/listings.

In addition, separate summary tables & listings will be produced for medical history possibly contributing to pulmonary diseases, and cardiovascular events.

### 2.3.4 Patient disposition

All randomly allocated patients by center will be summarized for all enrolled patients by Cohort using the FAS The number (%) of enrolled patients included in the FAS will be presented overall and by Cohort. The number (%) of screened, enrolled and not - enrolled patients and the reasons for screening failure will also be displayed. The number (%) of patients in the FAS who are still on treatment, who discontinued the study phases and the reason for discontinuation will be presented overall and by Cohort.

The following summaries will be provided (with % based on the total number of FAS patients):

- Number (%) of patients who were enrolled (based on data from IRT system)
- Number (%) of patients who were enrolled but not treated (based on DAR eCRF page not completed for any study medication component)
- Primary reason for not being treated (based on "End of Screening Phase" and "Withdrawal of Informed Consent(s)" eCRF pages)
- Number (%) of patients who were treated (based on DAR eCRF pages of each study medication completed with non-zero dose administered)
- Number (%) of patients who completed the study medication (based on the "Completion of Treatment disposition phase" Disposition eCRF page)
- Number (%) of patients who discontinued the study medication (based on the "End of Treatment Disposition" page)
- Primary reason for study medication phase discontinuation (based on the "End of Treatment Disposition" page)
- Number (%) of patients who have entered the safety follow-up (based on the "Completed/Discontinuation of Post-Treatment follow-up" Disposition eCRF page)
- Number (%) of patients who completed the safety follow-up (based on the "Completion of Post-Treatment follow-up" Disposition eCRF page)
- Number (%) of patients who discontinued the safety follow-up (based on the "Discontinuation of post-Treatment follow-up" Disposition eCRF page)
- Primary reason for safety follow-up discontinuation (based on the "Discontinuation of post-Treatment follow-up" Disposition eCRF page)

Safety follow-up will not be reported in the disposition summary for primary analyses timepoint (24 weeks).

#### 2.3.5 Protocol deviations

The number (%) of patients in all the analysis sets with CSR reportable protocol deviations will be tabulated by deviation category (as specified in the Study Specification Document) overall and by Cohort. All CSR reportable protocol deviations will be listed.

# 2.4 Treatments (study medication, rescue medication, concomitant therapies, compliance)

# 2.4.1 Duration of exposure to study medication

The safety set (SS) will be used for all summaries of study medication.

The duration of exposure will be summarized for each study cohort A, B and C. The dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity) will be summarized for each study cohort by descriptive statistics.

- The number of participants will be summarized for SS by study cohort.
- The number (%) of patients who have dose reductions or interruptions, and the reasons, will be summarized by cohort.
- Patient level listings of all doses administered on medication along with dose change reasons will be produced.
- Duration of exposure to study medication is considered by taking into account the duration of exposure of non-zero doses to the investigational drug or control.
- Time on treatment(weeks) = [(date of last administration of study medication) (date of first administration of study medication) (days with zero dose) + 1] / 7.
- Duration of exposure to study treatment (weeks) = [(date of last administration of study medication) (date of first administration of study medication) + 1] / 7.
- The date of last administration of study medication is defined in Section 2.1.1.
- Summary of duration of exposure of study medication will include categorical summaries based on intervals (<24 weeks, ≥24 weeks and < 48 weeks, ≥48 weeks and < 72 weeks, >=72 weeks) and continuous summaries (i.e., mean, standard deviation etc.).

#### **Cumulative dose**

Cumulative dose of a study medication is defined as the total dose given during the study medication exposure.

The **planned cumulative dose** for a study medication refers to the total planned dose as per the protocol up to the last date of study medication administration. The calculations for the three separate doses of study medication are:

- Cohort A (ABL001): 40 mg/administration × 2 (administration/day) × duration of exposure (days)
- Cohort B (ABL001): 80 mg/administration × 1 (administration/day) × duration of exposure (days)
- Cohort C (ABL001): 200 mg/administration × 2 (administration/day) × duration of exposure (days)

The **actual cumulative dose** refers to the total actual dose administered, over the duration for which the patient is on the study medication as documented in the DAR eCRF. It is the sum of the non-zero total daily doses recorded over the dosing period. For patients who did not take any drug the actual cumulative dose is by definition equal to zero. The actual cumulative dose will be summarized for each of the Cohort.

# Dose intensity and relative dose intensity

**Dose intensity** (DI) for patients with non-zero duration of exposure is defined as follows: DI (mg/day) = Actual cumulative dose (mg) / Duration of exposure to study treatment(days). For patients who did not take any drug the DI is by definition equal to zero.

#### **Planned dose intensity** (PDI) is defined as:

PDI (mg/day) = Planned cumulative dose (mg) / Duration of exposure to study treatment(days).

Relative dose intensity (RDI (%)) is defined as follows:

RDI (%) = [DI (mg/day) / PDI (mg/day)]\*100.

DI and RDI (%) will be summarized separately for all the three study Cohorts.

#### Dose changes, interruptions or permanent discontinuations

The number of patients, who have dose reductions, dose interruptions or permanent discontinuations, and the reasons, will be summarized separately for all the three study cohorts.

'Dose Reduced', 'Dose Interrupted' and 'Dose Permanently Discontinued' fields from the DAR eCRF pages will be used to determine the dose reductions, dose interruptions, and permanent discontinuations, respectively.

The corresponding fields, 'Reason for Dose Reduction', 'Reason for Dose Interruption and 'Reason for Permanent Discontinuation' will be used to summarize the reasons.

A dose change occurs when total daily dose is different from the most recently planned dose. For patients in Cohort A, there is only one planned dose, i.e., 40 mg b.i.d. For patients in Cohort B, there is only one planned dose, i.e., 80 mg/day QD. For patients in Cohort C, the initial planned dose is 200 mg b.i.d i.e., 400 mg/day.

For summarizing interruptions and reasons, multiple entries for interruption that are entered on consecutive days with different reasons will be counted as separate interruptions. However, if the reason is the same in the mentioned multiple entries on consecutive days, then it will be counted as one interruption.

**Reduction**: A dose reduction is where the actual total daily dose is lower than the most recently planned dose. Therefore, any dose reduction to correct a dosing error will not be considered a dose reduction. Only dose reduction is collected in the eCRF and will be summarized for the patient's data available.

#### 2.4.2 Prior, concomitant and post therapies/medication

### Prior antineoplastic therapy/medications

The number and percentage of patients who received any prior anti-neoplastic therapy /medications will be summarized by cohort and also for the lowest anatomical therapeutic classification (ATC) class and preferred term. Summaries will include total number of regimens.

Anti-neoplastic medications will be coded using the WHO Drug Dictionary (WHO-DD). Details regarding WHO-DD version will be included in the footnote in the tables/listings.

The above analyses will be performed using the SS.

# Post treatment anti-neoplastic therapy/medication

The number and percentage of patients who received any anti-neoplastic medication and/or therapy since discontinuation of study medication will be summarized by cohort for setting (e.g., adjuvant, metastatic, etc.) and for the lowest anatomical therapeutic classification (ATC) class and preferred term. Summaries will include total number of regimens, reason for initiation of new therapy, indication, route of administration and reason for discontinuation of therapy.

Anti-neoplastic medications will be coded using the WHO-DD. Details regarding WHO-DD version will be included in the footnote in the tables/listings.

The above analyses will be performed using the SS.

# **Prior and Concomitant therapies/Medications**

Prior and Concomitant therapies/medications are defined as all interventions (therapeutic treatments and procedures) other than the study medication administered to a patient coinciding with the study medication period. Prior therapies include medications (other than study drugs) and medical procedures started and ended prior to the start date of study medication. Concomitant therapies include medications (other than study drugs) and medical procedures starting on or after the start date of study medication but no later than 30 days after last dose of study medication or starting prior to the start date of study medication and continuing after the start date of study medication.

Prior and Concomitant therapies/medications will be coded using the World Health Organization (WHO) Drug Reference Listing (DRL) dictionary that employs the WHO ATC classification system and summarized by the lowest ATC class and PT using frequency counts and percentages. Surgical and medical procedures will be coded using MedDRA and summarized by SOC and PT. These summaries will include:

- Prior therapies/medications started and ended prior to the start date of study medication.
- Concomitant therapies/medications:
- 1. Therapies/medications starting on or after the start of study medication but no later than 30 days after last dose of study medication and
- 2. Therapies/medications starting prior to start of study medication and continuing after the start of study medication.

All prior & concomitant therapies/medications will be listed. Any concomitant therapies/medications starting and ending prior to the start of study medication or starting more than 30 days after the last date of study medication will be flagged in the listing. The safety set will be used for all concomitant therapies/medications' tables and listings.

# 2.5 Analysis of the primary objective

The primary objective is to evaluate safety profile of monotherapy asciminib in CML-CP in 3L and beyond for Cohorts A, and B. For all primary safety analyses, the Safety Set (SS) will be used, unless stated otherwise.

The variables for the primary analysis are incidence and severity of AEs and SAEs, changes in laboratory values and vital signs, incidence of notable ECG abnormalities.

## 2.5.1 Primary endpoint

The primary endpoint is to evaluate the safety profile of monotherapy asciminib (ABL001) with AEs, SAEs and laboratory studies' assessment during 24 weeks of therapy in CML-CP patients, for Cohorts A and B i.e., without T315I mutation status. All safety analyses will be based on the safety set (SS).

AE summaries will include all AEs occurring during on-treatment period. All AEs collected in the AE eCRF page will be listed along with the information collected on those AEs e.g., AE relationship to study drug, AE outcome, etc. AEs with start date outside of on-treatment period will be flagged in the listings.

AEs will be summarized by number and percentage of patients having at least one AE, having at least one AE in each primary system organ class (SOC) and for each preferred term (PT) using MedDRA coding. A patient with multiple occurrences of an AE will be counted only once in the respective AE category. A patient with multiple CTCAE grades for the same preferred term will be summarized under the maximum CTCAE grade recorded for the event. AE with missing CTCAE grade will be included in the 'All grades' column of the summary tables. Abnormal lab findings, vital signs and notable ECG abnormalities will also be summarized by cohort as explained in Safety analysis section 2.6.

# 2.5.2 Statistical hypothesis, model, and method of analysis

No formal hypothesis testing is planned for this study.

For all safety analyses, the safety set will be used.

#### 2.5.3 Handling of missing values

Missing data for measures of safety will not be imputed.

# 2.6 Safety analyses

All safety analyses will be based on the safety set (SS). All listings and tables will be presented by Cohort.

#### 2.6.1 Adverse events (AEs)

All the adverse events reported after administration of study drug to 30 days after the last date of drug to the patient are known as treatment emergent adverse events (TEAEs).

The summary tables for adverse events (AEs) will summarize only on-treatment events, with a start date during the on-treatment period (*treatment-emergent* AEs). In addition, a separate summary for death including on-treatment deaths will be provided. All AE will be listed and those collected during the on-treatment period (TEAE) will be flagged.

TEAEs will be summarized by number and percentage of patients having at least one AE in each primary system organ class (SOC) and for each preferred term (PT) using MedDRA coding. A patient with multiple occurrences of an AE will be counted only once in the respective AE category. A patient with multiple CTCAE grades for the same preferred term will be summarized under the maximum CTCAE grade recorded for the event. TEAE with missing CTCAE grade will be included in the 'All grades' column of the summary tables.

In TEAE summaries, the primary system organ class will be presented alphabetically, and the preferred terms will be sorted within primary SOC in descending frequency. The sorting order for the preferred term will be based on their frequency in the ABL001 arm Cohort A.

The following treatment emergent adverse event summaries will be produced by Cohort:

• Overview of TEAEs and deaths

- TEAEs by SOC and PT
- Summary by relationship
- Seriousness
- Leading to treatment discontinuation
- Leading to dose interruption/adjustment
- Requiring additional therapy and leading to fatal outcome

For posting to ClinTrial.gov and EudraCT, a summary table of on-treatment deaths and serious AEs and another summary table of non-serious AEs by treatment, both including occurrences (an occurrence is defined as >1 day between start and prior end date of record of same preferred term) and sorted by SOC and PT, will be presented as well.

All the adverse events will be graphically displayed by Cohorts using bar chart.

# 2.6.2 Adverse events of special interest / grouping of AEs

# **Data analysis of AESIs**

An adverse event of special interest (AESI) are defined as adverse events (serious or non-serious) which are of scientific and medical concern specific to compound ABL001 as mentioned in <u>Table 5-5</u>. For which ongoing monitoring and rapid communication by the investigator to the sponsor may be appropriate. Such events may require further investigation in order to characterize and understand them.

Adverse events of special interest are defined on the basis of an ongoing review of the safety data. The latest approved version of CRS prior to the respective database lock will be used.

For each specified AESI, number and percentage of patients with at least one event of the AESI occurring during the on-treatment period will be summarized.

Summaries of these AESIs will be provided by cohort. If sufficient number of events occurred, analysis of time to first occurrence will be applied.

A listing of all grouping levels down to the MedDRA PTs used to define each AESI will be generated.

#### 2.6.3 Deaths

Separate summaries for on-treatment / TEAE and all deaths will be produced by system organ class and preferred term, by cohort.

All deaths will be listed, where on treatment deaths will be flagged. A separate listing of deaths prior to starting treatment will be provided for all screened patients.

#### 2.6.4 Laboratory data

Grading of laboratory values will be assigned programmatically as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The calculation of CTCAE grades will be based on the observed laboratory values only, clinical assessments will not be taken into account. CTCAE Grade 0 will be assigned for all non-missing values not graded as 1 or higher. Grade 5 will not be used. Details of CTCAE grading and imputation rules are presented in Appendix 5.3.

For laboratory tests where grades are not defined by CTCAE v5.0, results will be categorized as low/normal/high based on laboratory normal ranges.

On analyzing laboratory, data from all sources (central and local laboratories) will be combined. The summaries will include all assessments available for the laboratory parameter collected no later than 30 days after the last study medication administration date.

The following summaries will be produced separately for hematology and biochemistry laboratory data (by laboratory parameter and cohort):

- Worst post-baseline CTCAE grade (regardless of the baseline status). Each patient will be counted only for the worst grade observed post-baseline in the on-treatment period.
- Shift tables to compare baseline CTCAE grades to the worst on-treatment grade for laboratory tests where grades are not defined by CTCAE v5.0
- Shift tables using the low/normal/high/ (low and high) (or project specific) classification to compare baseline to the worst on-treatment value.
- Newly or worsening laboratory abnormalities will be summarized, separately.

The following listings will be produced separately for hematology and biochemistry for the laboratory data:

- Listings of all laboratory data, with corresponding CTCAE grades and classification relative to the laboratory normal range. Lab data collected during the post-treatment period with corresponding CTCAE v5 grades will be flagged.
- Listing of all CTCAE grade 3 or 4 laboratory toxicities
- Box plot(s) for all laboratory parameters over time will be plotted and displayed by Cohort.

#### 2.6.5 Other safety data

#### 2.6.5.1 ECG and cardiac imaging data

12-lead ECGs including PR, QRS, QT, QTcF and RR intervals will be obtained centrally for each patient during the study. ECG data will be read and interpreted centrally.

Absolute values/change from baseline will be summarized over time. As appropriate, the number and percent of patients will be tabulated by category. In addition, a listing of patients with at least one notable ECG value will be produced.

#### Data handling

The average of the triplicate ECG parameters at each time point will be used in the analyses.

# Data analysis

The number and percentage of patients with notable ECG values will be presented by Cohort. Notable values are defined below:

- QT, QTcF
  - New value of > 480 and  $\le 500$  ms
  - New value of > 500 ms
- HR
  - Increase from baseline >25% and to a value > 100 bpm
  - Decrease from baseline >25% and to a value < 50 bpm

- PR
  - Increase from baseline >25% and to a value > 200 ms
  - New value of > 200 ms
- ORS
  - Increase from baseline >25% and to a value > 120 ms
  - New values of QRS > 120 ms

A listing of only the patients with notable ECG values will be produced. In the listing the assessments collected during the on-treatment period will be flagged.

### 2.6.5.2 Vital signs

Data on vital signs will be tabulated and summarized descriptively as follows:

• Number and percentage of patients who shift from non-notable at baseline to notable post- baseline. Also, bar chart with 95% CI will be presented for the notable changes.

The number and percentage of patients with notable vital sign values (high/low) in systolic blood pressure, diastolic blood pressure, pulse rate, weight and temperature will be presented by Cohort.

A listing of notable vital sign values will be produced. In the listing, the assessments collected outside of on-treatment period will be flagged.

# 2.6.5.3 Cardiovascular and Pulmonary risk factor assessment

Prior to random allocation of patients to cohort and at the end of treatment, cardiovascular risk factors collected will be listed by cohort.

Prior to random allocation of patients to cohort and at Week 20, pulmonary function tests including assessment of the lung volumes FEV1, FVC, FEV1/FVC, TLC, VC and DLCO will be performed, if clinically indicated. A listing will be presented by cohort.



# 2.7 Analysis of the key secondary objective

Not applicable

# 2.8 Analysis of the secondary objective(s)

The secondary objective(s) of the study are:

- To estimate the rate of hematologic and molecular responses at specific time points for
- Cohort A, B and C
- Rate of CHR, MR2, MMR, MR4, MR4.5 in 12, 24, 48, 72 weeks of therapy
- To estimate time to hematologic and molecular response
- Time to CHR, MR2, MR4, MR4.5 in 12, 24, 48, 72 weeks of therapy

- To evaluate the duration of hematologic and molecular response
- Duration of MR1, MR2, MMR, MR4 and MR4.5
- To evaluate Progression Free Survival (PFS)
- To evaluate Overall Survival (OS)

#### 2.8.1 Secondary safety endpoints

The secondary safety endpoints are:

• AEs, SAEs and laboratory evaluation for Cohort A, Cohort B and Cohort C, by 48, 72 weeks

All secondary safety analysis will be performed similar to the above primary safety analysis using Safety set (SS) by 48, 72 weeks. Additionally, a separate safety summary up to 24 weeks will be provided for Cohort C.

# 2.8.2 Secondary efficacy endpoints

The secondary efficacy endpoints are:

- Rate of CHR, MR2, MMR, by 12, 24, 48, 72 weeks of therapy
- Rate of MR4, MR4.5 by 24, 48, 72 weeks of therapy
- Time to CHR, MR2, MMR, MR4, MR4.5
- Duration of CHR, MR2, MMR, MR4 and MR4.5
- PFS during 24, 48 and 72 weeks
- OS during 24, 48 and 72 weeks

For all secondary efficacy analyses, the Full Analysis Set (FAS) will be used, unless stated otherwise.

For secondary efficacy analysis, proportion of patients achieving the response levels will be presented together with an exact 95% Clopper-Pearson confidence interval. For time to event and duration, PFS & OS, median, 25<sup>th</sup> percentile & 75<sup>th</sup> percentile will be reported along with their respective 95% Confidence Interval.

# Rate of CHR, MR2, MMR, by 12, 24, 48, 72 weeks of therapy and Rate of MR4 & MR4.5 by 24, 48, 72 weeks of therapy

- The rate of Complete Hematologic Response (CHR) by 12, 24, 48 and 72 weeks. CHR is defined as all of the following present for  $\geq 4$  weeks:
  - WBC count  $< 10 \times 10^9/L$
  - Platelet count < 450 x 10<sup>9</sup>/L
  - Basophils < 5%
  - No blasts and promyelocytes in peripheral blood
  - Myelocytes + metamyelocytes < 5% in peripheral blood
  - No evidence of extramedullary disease, including spleen and liver
- The rate of **molecular response (MR2)** by 12, 24, 48 and 72 weeks after the start of first study medication. **MR2** is defined as  $\geq 2$  log reduction of BCR-ABL transcript from standardized baseline or  $\leq 1\%$  BCR-ABL/ABL % by international scale, measured by real-time quantitative PCR (RQ-PCR).

- The rate of **major molecular response (MMR)** by 12, 24, 48 and 72 weeks after the start of first study medication. MMR is defined as  $\geq 3$  log reduction of BCR-ABL transcript from standardized baseline or  $\leq 0.1\%$  BCR-ABL/ABL % by international scale, measured by real-time quantitative PCR (RQ-PCR).
- The rate of **molecular response (MR4)** by 24, 48 and 72 weeks after the start of first study medication. **MR4** is defined as  $\geq$  4 log reduction of BCR-ABL transcript from standardized baseline or  $\leq$  0.01% BCR-ABL/ABL % by international scale, measured by real-time quantitative PCR (RQ-PCR).
- The rate of the **molecular response (MR4.5)** by 24, 48 and 72 weeks after the start of first study medication. **MR4.5** is defined as  $\geq$  4.5 log reduction of BCR-ABL transcript from standardized baseline or  $\leq$  0.0032% BCR-ABL/ABL % by international scale, measured by real-time quantitative PCR (RQ-PCR).

For rate of MR2, MMR, MR4, MR4.5 by any pre-specified time point patients will be consider as responder if he/she achieve the particular response at least once by the specific timepoint. If patient discontinuing the treatment prior to a specific time point due to any reason and not achieved the particular response before the discontinuation will be considered as non-responder.

For each time point, the proportion of patients achieving the specific response levels will be presented together with an exact 95% Clopper-Pearson confidence interval by cohort. The rates over time will be displayed graphically using the Bar Charts with 95% C.I. as whiskers.

**Note:** Patient(s) who have reported for molecular response(s) at baseline will not be included in time to event analyses.

### Time to CHR, MR2, MR4, MR4.5 in 72 weeks of therapy

Time to achieving a response level is defined as the time from the date of the first dose of study medication to the first documented achievement of a response level.

Time to achieve a specific response level will be analyzed using the Kaplan-Meier Product- Limit method. Patients who are known to be without achieving that response level will be censored at the last molecular & hematologic assessment.

The estimated cumulative incidence rates and 95% confidence intervals at 12, 24, 48 and 72 weeks will be presented. The cumulative incidence curve will be plotted. , if applicable. The analyses will be performed using FAS by cohort.

For patients in the FAS who have not experienced any molecular and/or hematologic response, the time will be censored as follows in the Kaplan-Meier analysis:

- If a patient does not achieve the specified response before the cut-off date for the analysis, censoring time will be the last molecular assessment (PCR) date on treatment prior to the cut-off date or the EoT visit, whichever comes first.
- If a patient discontinues study treatment prior to achieving a response for a reason other than disease progression or death, then the patient will be censored at the last molecular assessment (PCR) date on treatment prior to the cut-off date or the EoT visit, whichever comes first.

• If a patient discontinues study treatment prior to achieving a response due to progression or death, then the censoring time will be set to the longest follow-up time in the treatment group, that is, consider the response is impossible to reach.

In case no on-treatment response assessment was performed, the patient will be censored at day 1.

## Duration of CHR, MR2, MMR, MR4 and MR4.5

Duration of Response (DOR) is the time from the date of the first documented molecular (MR2, MMR, MR4, MR4.5) or Hematologic (CHR) response to the date of first documented loss of that response or death due to any cause or progression to AP/BC, whichever occurs first.

The start date is the date of first documented response and the end date is defined as the date of the first documented loss of that response or death due to any cause or progression to AP/BC. Participants continuing without that event will be censored at the date of their last adequate molecular of hematologic response assessment.

DOR for each response level will be analyzed using the Kaplan-Meier Product-Limit method.

Estimates of DOR at specific timepoint and the 25th, median and 75th percentile of the DOR and their 95% confidence intervals will be provided, if applicable.

# 2.8.1.1 Other secondary efficacy endpoints

**Progression-Free-Survival (PFS)** is defined as time from the first dose of study medication to disease progression to AP/BC or death due to any cause, whichever occurs first during 24,48 and 72 weeks.

For patients without progression, the patient will be censored at the last molecular assessment date the patient was known to be alive and without progression (on or before the cut-off date).

PFS will be analyzed using the Kaplan-Meier Product-Limit method. Patients who do not progress will be censored at the last adequate assessment. Estimates of the 25th, median and 75th percentile of the PFS and their 95% confidence intervals will be provided, if applicable.

**Overall survival (OS)** is defined as the time from the first dose of study medication to death due to any cause during 24, 48 weeks and 72 weeks during study.

If a patient is not known to have died, then OS will be censored at the latest date the patient was known to be alive (on or before the cut-off date). All deaths will be taken into account whatever the death occurred, i.e., even after interruptions, or discontinuation of study medication due to any reason.

OS will be analyzed using the Kaplan-Meier Product-Limit method. Patients who do not progress will be censored at the last adequate assessment. Estimates of the 25th, median and 75th percentile of the OS and their 95% confidence intervals will be provided, if applicable.

# 2.8.3 Handling of missing values/censoring/discontinuations

## MMR rates by specific time points:

Patients without any documented response for which an evaluable response assessment was never provided will be considered as non-responders for the period of time up to that time point.

**Molecular response category by specific time points**: The category "Missing" will be assigned to patients for whom an evaluable response assessment was never provided.

**Time to MMR**: For patients in the FAS who have not experienced any MMR, the time will be censored as follows in the Kaplan-Meier analysis:

If a patient does not achieve the specified response before the cut-off date for the analysis, censoring time will be the last molecular assessment (PCR) date on treatment prior to the cut-off date or the EoT visit, whichever comes first.

If a patient discontinues study treatment prior to achieving a response for a reason other than disease progression or death, then the patient will be censored at the last molecular assessment (PCR) date on treatment prior to the cut-off date or the EoT visit, whichever comes first.

If a patient discontinues study treatment prior to achieving a response due to progression or death, then the censoring time will be set to the longest follow-up time in the treatment group, that is, consider the response is impossible to reach.

In case no on-treatment response assessment was performed, the patient will be censored at day 1.

**Duration of MMR**: For patients who have not experienced any event (loss of MMR, progression to AP/BC, or CML-related death), the duration will be censored at the last molecular assessment (PCR) date on treatment.

**PFS**: For patients who have not experienced protocol defined event (disease progression to AP/BC or death from any cause), the patients will be censored at the date of last study assessment (PCR, cytogenetic, hematologic or extramedullary) before the cut-off date.

**OS**: Patients who are alive at the time of the analysis data cutoff date will be censored at the date of last contact (see Section 2.1.1) before the cut-off date.

#### 2.8.4 Statistical hypothesis, model, and method of analysis

There is no formal hypothesis to test in this study.







# 2.10 Interim analysis

As the primary time point is by 24 weeks, the primary analysis will be an interim analysis. The primary analysis will be performed when the last patient completes 24 weeks of treatment or discontinues early.

As appropriate, annual interim analyses will be planned for publication or any regulatory purpose. No formal interim analysis will be performed. Only summary statistics will be provided.

Final Analysis will be performed when the last patient completes 72 weeks or discontinues early. A final CSR will be written.

# 3 Sample size calculation

This is an open label, three-cohort study to assess safety and efficacy of study of asciminib (ABL001) monotherapy in patients with chronic myeloid leukemia in chronic phase (CML-CP) previously treated with at least 2 prior TKIs (tyrosine kinase inhibitors) and CML-CP patients harboring the T315I mutation previously treated with at least 1 prior TKIs.

For all CML-CP with the exception of those harboring the T315I mutation, there will be random allocation of patients to eliminate selection bias at the time of cohort allocation. Those patients will be assigned to either Cohort A consisting of asciminib 40 mg BID patients or Cohort B consisting of asciminib 80 mg QD. For CML-CP patients harboring the T315I mutation, they will be assigned to Cohort C with asciminib 200 mg BID, which is the dose required for that patient population. It is worthwhile mentioning that random allocation of patients in cohorts A and B will be pursued for patient selection only. The study is not powered to show differences in Primary and Secondary endpoints between study cohorts.

Primary objective of the study is to assess safety profile of this combination drug during 24 weeks for all cohort patients.

A sample size of 40 evaluable patients for Cohort A is estimated based on a two- sided 95% confidence interval for an incidence rate of an AE using the large sample normal approximation that will extend 0.12 from the observed incidence rate of an AE (precision or margin of error of 12%) for an expected incidence rate of 18%. Considering drop-out rate of 10%, approximately 45 patients will be enrolled for safety assessment for the Cohort A of this study.

Retaining the same assumptions, approximately 45 patients will also be enrolled for Cohort B. Additionally for Cohort C, approximately 25 patients will be enrolled.

Thus, approximately total 115 (45+45+25=115) patients will be enrolled for Cohort A (n1=45) and Cohort B (n2=45) and for Cohort C (n3=25) of the study.

# 4 Change to protocol specified analyses

No change to the protocol specified analysis has been made.

# 5 Appendix

# 5.1 Imputation rules

# 5.1.1 Study drug

The following rules should be used for the imputation of the dose end date for a given study medication component.

<u>Scenario 1</u>: If the dose end date is completely missing and there is <u>no EOT page</u> and <u>no death</u> <u>date</u>, the patient is considered as on-going:

The patient should be treated as on-going and the cut-off date should be used as the dose end date.

<u>Scenario 2</u>: If the dose end date is completely or partially missing and the <u>EOT page</u> is available:

- Case 1: The dose end date is completely missing, and the EOT completion date is complete, then this latter date should be used.
- Case 2: Only Year(yyyy) of the dose end date is available and yyyy < the year of EOT date: Use Dec31yyyy
- Case 3: Only Year(yyyy) of the dose end date is available and yyyy = the year of EOT date: Use EOT date
- Case 4: Both Year(yyyy) and Month (mm) are available for dose end date, and yyyy = the year of EOT date and mm < the month of EOT date:

  Use last day of the Month (mm)
- All other cases should be considered as a data issue and the statistician should contact the data manager of the study.
- After imputation, compare the imputed date with start date of treatment, if the <u>imputed date is <</u> start date of treatment:
- Use the treatment start date

Patients with missing start dates are to be considered missing for all study medication component related calculations and no imputation will be made. If start date is missing then end-date should not be imputed.

#### 5.1.2 AE, ConMeds and safety assessment date imputation

The imputations specified in this section are only used for analyses of time to and duration of AEs and concomitant medications.

Table 5-1 Imputation of start dates (AE, CM) and assessments (LB, EG, VS)

| Missing<br>Element | Rule |
|---|---|
| day, month, and year | No imputation will be done for completely missing dates |
| day, month | <ul> <li>If available year = year of study medication study medication start date then <ul> <li>If stop date contains a full date and stop date is earlier than study medication study medication start date then set start date = 01JanYYYY</li> <li>Else set start date = study medication study medication start date.</li> </ul> </li> <li>If available year &gt; year of study medication study medication start date then 01JanYYYY</li> <li>If available year &lt; year of study medication study medication start date then 01JulYYYY</li> </ul> |
| Day | <ul> <li>If available month and year = month and year of study medication study medication start date then <ul> <li>If stop date contains a full date and stop date is earlier than study medication study medication start date then set start date= 01MONYYYY.</li> <li>Else set start date = study medication study medication start date.</li> </ul> </li> <li>If available month and year &gt; month and year of study medication study medication start date then 01MONYYYY</li> <li>If available month and year &lt; month year of study medication study medication start date then 15MONYYYY</li> </ul> |

Table 5-2 Imputation of end dates (AE, CM)

| Missing<br>Element | Rule (*=last treatment date plus 30 days not > (death date, cut-off date, withdrawal of consent date)) |
|---|---|
| day, month,<br>and year | Completely missing end dates (incl. ongoing events) will be imputed by the end date of the on-treatment period* |
| day, month | • If partial end date contains year only, set end date = earliest of 31DecYYYY or end date of the on-treatment period * |
| Day | • If partial end date contains month and year, set end date = earliest of last day of the month or end date of the on-treatment period* |

Any AEs and ConMeds with partial/missing dates will be displayed as such in the data listings.

Any AEs and ConMeds which are continuing as per data cut-off will be shown as 'ongoing' rather than the end date provided.

#### 5.1.2.1 Other imputations

### Incomplete date of initial diagnosis of cancer

Completely missing dates will not be imputed. Partial dates of diagnosis will be compared to the treatment start date.

- If DIAG year < study treatment start date year and DIAG month is missing, the imputed DIAG date is set to the mid-year point (01JULYYYY).
- Else if DIAG month is not missing, the imputed DIAG date is set to the mid-month point(15MONYYYY).
- If DIAG year = study treatment start date year and (DIAG month is missing OR DIAG month is equal to study treatment start month), the imputed DIAG date is set to one day before study treatment start date.

# 5.2 AEs coding/grading

Adverse events are coded using the latest available version of Medical dictionary for regulatory activities (MedDRA) terminology.

AEs will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

The CTCAE represents a comprehensive grading system for reporting the acute and late effects of cancer treatments. CTCAE grading is by definition a 5-point scale generally corresponding to mild, moderate, severe, life threatening, and death. This grading system inherently places a value on the importance of an event, although there is not necessarily proportionality among grades (a grade 2 is not necessarily twice as bad as a grade 1).

# 5.3 Laboratory parameters derivations

Grade categorization of lab values will be assigned programmatically as per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The calculation of CTCAE grades will be based on the observed laboratory values only, clinical assessments will not be taken into account. The criteria to assign CTCAE grades are given in Novartis internal criteria for CTCAE grading of laboratory parameters (embedded below). The latest available version of the document based on the underlying CTCAE version v5.0 at the time of analysis will be used. For laboratory tests where grades are not defined by CTCAE v5.0, results will be graded by the low/normal/high (or other project-specific ranges, if more suitable) classifications based on laboratory normal ranges.

A severity grade of 0 will be assigned for all non-missing lab values not graded as 1 or higher. Grade 5 will not be used. For laboratory tests that are graded for both low and

high values, summaries will be done separately and labelled by direction, e.g., sodium will be summarized as hyponatremia and hypernatremia.



#### Imputation Rules

CTCAE grading for blood differentials is based on absolute values. However, this data may not be reported as absolute counts but rather as percentage of white blood cells (WBC).

If laboratory values are provided as '<X' (i.e. below limit of detection) or '>X', prior to conversion of laboratory values to SI unit, these numeric values are set to X.

The following rules will be applied to derive the WBC differential counts when only percentages are available for a xxx differential

xxx count = (WBC count) \* (xxx %value / 100)

The following rules will be applied to derive the WBC differential percentages when only differential counts are available for a xxx differential

xxx%value =  $(xxx count \times 100) / WBC count$ 

Further derivation of laboratory parameters might be required for CTCAE grading. For instance, corrected calcium can be derived using the reported total calcium value and albumin at the same assessment using the following formula:

Corrected Calcium (mg/dL) = Calcium (mg/dL) - 0.8 [Albumin (g/dL)-4]

In order to apply the above formula, albumin values in g/L will be converted to g/dL by multiplying by 0.1 and calcium values in mmol/L will be converted to mg/dL by dividing by 0.2495. For calculation of laboratory CTCAE grades 0 and 1, the normal range for derived corrected calcium is set to the same limits (in mg/dL) as for calcium.

CTCAE grades for the derived absolute WBC differential counts (neutrophils, lymphocytes) and corrected calcium will be assigned as described above for grading.

# 5.3.1 Derivation of PCR results and loss of response(s)

Scaling towards an international standard will be performed for all molecular results using laboratory specific conversion factors. In this process, the raw ratio between BCR-ABL and the control gene ABL is calculated and multiplied by the lab -specific conversion factor ([Branford and Hughes 2006]). Therefore, using the international unit, the BCR-ABL ratio will be presented in %. The MRDx assay using PAXgene TM Blood RNA tubes from MMD laboratory will be used in this study. The lab conversion factor for this assay is 1.1.

The BCR-ABL ratio in IS % is calculated by multiplying the raw BCR-ABL ratio with the lab-specific conversion factor and then by 100:

BCR-ABL ratio (in %) = (BCR-ABL / ABL) \* conversion factor \* 100

For consistency with elsewhere reported molecular response rates, the result may be expressed also as log-reduction. This is defined as the following:

BCR-ABL Log-Reduction = -log<sub>10</sub> (BCR-ABL ratio in %)

For example,  $-\log_{10}(0.001) = 3 \log reduction$  for a ratio of 0.1%.

The following binary variables will be used when molecular response is reported.

Table 5-3 Response categories for molecular response

| MR (Molecular Response) | | BCR-ABL ratio (%) | Log-reduction category |
|-------------------------|-----|-------------------|------------------------|
| MMR | Yes | ≤ 0.1% | ≥ 3-log reduction |
| IVIIVIK | No | > 0.1% | < 3-log reduction |
| | Yes | ≤ 1% | $\geq$ 2 log reduction |
| MR2 | No | > 1% | < 2 log reduction |
| | Yes | ≤ 0.01% | ≥ 4 log reduction |
| MR4 | No | > 0.01% | < 4 log reduction |
| MR4.5 | Yes | ≤ 0.0032% | ≥ 4.5-log reduction |
| WIK4.3 | No | > 0.0032% | < 4.5-log reduction |

#### **Loss of Responses**

Loss of MR2 is defined as increase of BCR-ABL/ABL to > 1% by international scale (IS). BCR-ABL less than 1% according to the IS can be regarded as an equivalent to CCyR. Loss of MR2 must be confirmed by subsequent sample analysis within 4 to 6 weeks.

Loss of MMR is defined as increase of BCR-ABL/ABL to > 0.1% by international scale (IS) in association with a  $\ge 5$ -fold rise in BCR-ABL from the lowest value achieved on study treatment and replicated by a second analysis of the same sample. Loss of MMR must be confirmed by subsequent sample analysis within 4 to 6 weeks showing loss of MMR associated with a  $\ge 5$ -fold rise in BCR-ABL from the lowest value achieved on study treatment, unless it is associated with confirmed loss of CHR to AP/BC or CML-related death.

# 5.4 Listing of AESIs

All the adverse event of special interest (AESI) that are of scientific and medical concern specific to compound ABL001, collected from previous trials are mentioned below with Preferred Term (PT) and system Organ Class (SOC) in <u>Table 5-5</u>.

Table 5-4 List of AESIs reported for ABL001(Asciminib)

| Preferred Tem | System Organ Class |
|---|---|
| Pancreatic toxicity | Gastrointestinal disorders |
| Hemorrhage | Vascular disorders |
| Edema and fluid retention | General disorders and administration site conditions |
| Hepatotoxicity (including laboratory terms) | Hepatobiliary disorders |
| Myelosuppression (Leucopenia) | Blood and lymphatic system disorders |
| Hypersensitivity | Immune system disorders |
| Hepatotoxicity (clinical events) | Hepatobiliary disorders |
| GI toxicity | Gastrointestinal disorders |
| Pancreatic toxicity (clinical events) | Gastrointestinal disorders |
| Myelosuppression (Thrombocytopenia) | Blood and lymphatic system disorders |
| Hepatotoxicity (including laboratory terms) | Hepatobiliary disorders |
| QTc prolongation | Cardiac disorders |
| Ischemic heart and CNS conditions | Vascular disorders |
| Hepatotoxicity (including laboratory terms) | Hepatobiliary disorders |
| Hepatotoxicity (including laboratory terms) | Hepatobiliary disorders |
| Cardiac failure (clinical events) | Cardiac disorders |
| Phototoxicity | Skin and subcutaneous tissue disorders |
| Myelosuppression (cytopenias affecting more than one lineage) | Blood and lymphatic system disorders |
| Myelosuppression (Erythropenia) | Blood and lymphatic system disorders |
| Ischemic heart and CNS conditions | Vascular disorders |
| Reproductive toxicity | Reproductive system and breast disorders |
| Hepatitis B virus reactivation | Infections and infestations |
| Hepatotoxicity (clinical events) | Hepatobiliary disorders |

### 6 Reference

- 1. Armitage P, McPherson CK and Rowe BC (1969). Repeated significance tests on accumulating data. J.R. Statist. Soc. A, 132, 232-244.
- 2. Baccarani M, Deininger DW, Rosti G, et al (2013). European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013. Blood; 122(6):872-84.
- 3. Branford S, Hughes T (2006) Diagnosis and monitoring of chronic myeloid leukemia by qualitative and quantitative RT-PCR. Methods Mol Med; 125:69-92.
- 4. Brookmeyer R and Crowley J (1982). A Confidence Interval for the Median Survival Time. Biometrics, 38, 29 41.
- 5. Clopper CJ and Pearson ES (1934). The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrical, 26, 404-413.
- 6. Collet D (1994). Modelling survival data in medical research. London, Chapman & Hall.
- 7. Gambacorti-Passerini C, Brümmendorf TH, Kim DW, et al (2014). Bosutinib efficacy and safety in chronic phase chronic myeloid leukemia after imatinib resistance or intolerance: Minimum 24-month follow-up. Am J Hematol; 89(7):732-42.
- 8. García-Gutiérrez V, Martinez-Trillos A, Lopez Lorenzo JL, et al (2015). Bosutinib shows low cross intolerance, in chronic myeloid leukemia patients treated in fourth line. Results of the Spanish compassionate use program. Am J Hematol; 90(5):429-33.
- 9. Khoury HJ, Cortes JE, Kantarjian HM, et al (2012). Bosutinib is active in chronic phase chronic myeloid leukemia after imatinib and dasatinib and/or nilotinib therapy failure. Blood; 119(15):3403-12.
- 10. Mantel, N. and Joseph L Fleisś (1980). Minimum expected cell size requirements for the Mantel-Haenszel one degree-of-freedom Chi-Square Test and a related rapid procedure. American Journal of Epidemiology, 112, 129-134.
- 11. European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013; Prepublished online 2013 Jun 26. doi: 10.1182/blood-2013-05-501569; PMCID: PMC4915804; PMID: 23803709